CLINICAL TRIAL: NCT06125158
Title: Study on the Effect of Hip Strength Training and Neuromuscular Electrical Stimulation on the Intervention of Functional Ankle Instability of Sport
Brief Title: Effects of Hip Strength Training and Neuromuscular Electrical Stimulation on Functional Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin University of Sport (Other)
Responsible Party: Principal Investigator, Yanhua, Guo, student enrolled in a master's program, Tianjin University of Sport
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TianjinSport
Record Dates: First submitted 2023-11-05; First posted 2023-11-09 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Ankle Injuries and Disorders
MeSH Terms: conditions — Ankle Injuries; Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): Participants in this group will receive conventional ankle interventions including ankle strength training and balance training. All treatments target the affected lower extremity for 40 minutes per session, once per day, 3 days per week for 6 weeks.
  Interventions: Procedure: Conventional ankle training
- Experimental Group A (Experimental): Participants in this group will be asked to perform conventional ankle training and hip strength training. The conventional ankle training routine for this group will have the same movements as the control group, but the volume of training will be half that of the control group, and the duration of training will be 20 min/session. Hip strength training will consist of elastic band resistance exercises, forward step-up and lateral step-up for 20 min/session. All treatments target the affected lower extremity for 40 minutes per session, once per day, 3 days per week for 6 weeks.
  Interventions: Procedure: Conventional ankle training; Procedure: Hip strength training
- Experimental Group B (Experimental): Participants in this group will be asked to perform conventional ankle training and neuromuscular electrical stimulation. The conventional ankle training routine for this group will have the same movements as the control group, but the volume of training will be half that of the control group, and the duration of training will be 20 min/session. Neuromuscular electrical stimulation aims to stimulate the gluteus maximus and gluteus mediums muscles of the affected lower limb. The researcher chose the "Neuromuscular Electrical Stimulation 1" mode for the treatment prescription (this prescription can output a variety of waveforms with frequencies varying continuously from 1 to 100 Hz to stimulate the target muscles alternately, effectively preventing muscle fatigue caused by a single stimulation) and set the stimulation time to 20 min per session. All treatments target the affected lower extremity for 40 minutes per session, once per day, 3 days per week for 6 weeks.
  Interventions: Procedure: Conventional ankle training; Procedure: Neuromuscular electrical stimulation

INTERVENTIONS:
Procedure: Conventional ankle training — The program included ankle elastic band resistance training and balance training, in which the elastic band resistance training required subjects to complete resistance training in ankle plantarflexion, dorsiflexion, inversion and eversion directions with the help of elastic bands; and the balance training required subjects to complete the movements of standing with eyes open, standing with eyes closed, and throwing and catching the ball on flat ground and BOSU ball.
Procedure: Hip strength training — Hip strength training required subjects to complete resistance training in hip abduction and posterior extension, anterior step-up and lateral step-up exercises with the help of elastic bands.
  Arms: Experimental Group A
Procedure: Neuromuscular electrical stimulation — Neuromuscular electrical stimulation of the gluteus mediums and gluteus maximus muscles of the affected side was carried out using the TB6807 low-frequency therapeutic instrument (with prescription for neuromuscular electrical stimulation) manufactured by China Tangbang Science and Technology Company.
  Arms: Experimental Group B

SUMMARY:
The goal of this clinical trial is to compare the effects of two methods of elevating hip muscle strength on functional ankle instability(FAI). . The main question[s] it aims to answer are:

* Whether hip strength training and neuromuscular electrical stimulation of the gluteal muscles, respectively, based on conventional ankle training improves dysfunction in patients with FAI?
* Is there a difference in the efficacy of the above two interventions for FAI?

DETAILED DESCRIPTION:
Participants will be randomly divided into 3 groups (Experimental Group A, Experimental Group B and Control Group) to receive the intervention for 6 weeks. The Control Group will undergo conventional ankle interventions such as peri-ankle muscle strength training and ankle balance training; Experimental Group A will undergo hip muscle strength training based on the conventional training; and Experimental Group B will perform neuromuscular electrical stimulation of hip abductors and hip extensors based on the conventional training. Researchers will compare the three groups to see changes in hip muscle strength, lower extremity muscle activation, ankle muscle strength, proprioception, dynamic and static balance, and self-reported ankle function.

ELIGIBILITY:
Inclusion Criteria:

* History of at least one acute ankle sprain one year ago, accompanied by symptoms such as pain, swelling, and inability to participate in daily activities for more than one day.
* Unilateral ankle sprains and or instability felt at least twice during the past year.
* Last ankle sprain occurred greater than or equal to 1 month from the start of the experiment.
* Cumberland Ankle Instability Tool (CAIT) score less than or equal to 27 points,
* The results of Medial Talar Tilt Test and Anterior Draw Test are negative.
* Body Mass Index （BMI）ranges from 18 to 25.

Exclusion Criteria:

* History of lower extremity surgery or fracture.
* History of brain injury or neurological disorders.
* Acute injury to musculoskeletal structures of other joints of the lower extremities within 1 month, affecting joint integrity and function.
* Participated in lower extremity rehabilitation or systematic athletic training after injury.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2023-10-18 (Actual); Primary Completion 2023-12-02 (Actual); Study Completion 2023-12-23 (Actual)

PRIMARY OUTCOMES:
Cumberland Ankle Instability Tool (CAIT) score | Subjects were asked to test 1 time for 10 min before and after the intervention.
  Using the CAIT score reflects the participant's subjective level of perceived stability of the ankle joint. The questionnaire contains 9 questions related to ankle function, mainly about ankle stability, pain and ankle sprains during daily activities, such as walking, running, descending stairs, and standing on one or two legs, with scores ranging from 0 to 30. The higher the score, the better the ankle stability.
Dynamic and static balance | Subjects were asked to test 1 time for 20 min before and after the intervention.
  The Tecnobody PK254P Balance Tester was used to perform static postural stability tests and dynamic postural stability tests to assess the subject's static and dynamic balance abilities. Static Postural Stability Test and Dynamic Postural Stability Test to assess the static and dynamic balance ability of the subjects. Static balance was measured by the pre The static balance ability was measured by the standard deviation in the forward and backward directions, the standard deviation in the left and right directions, the area of the movement ellipse and the circumference of the movement trajectory. The static balance ability was measured by the total stability index, anterior-posterior axis stability index, and left-right axis stability index.
Muscle activation | Subjects were asked to test 1 time for 40 min before and after the intervention.
  The electromyographic signals of gluteus medius, gluteus maximus, tibialis anterior, peroneus longus and gastrocnemius were collected by Noraxon ultium wireless surface electromyography to analyze the total amount of discharges of the motor units of the target muscles when the target muscles were involved in the activity, so as to reflect the degree of activation of the motor units of the target muscles in the course of the exercise. The test index is the Root Mean Square (RMS) of the target muscles before and after the landing moment of the single-leg vertical jump test.
Joint position sense | Subjects were asked to test 1 time for 20 min before and after the intervention.
  Plantarflexion, dorsiflexion, inversion and eversion joint positional perception tests in active mode at the affected ankle joint were performed using the Humac Norm Multi-Joint Isokinetic Test and Training System to assess the subject's proprioception. Absolute Errors (AE) between the values of the active inversion and active valgus position sense tests and the values requested by the tester were measured.
Hip isometric strength | Subjects were asked to test 1 time for 20 min before and after the intervention.
  The Humac Norm model multi-joint isokinetic testing apparatus was used to perform hip abductor and extensor strength on the affected side in order to assess the subject's hip abductor and extensor strength. Peak Torque (PT), Relative Peak Torque to Body Weight (PT/BW), and Total Work (TW) were measured during centripetal contraction at 60°/s and 180°/s angular velocities.
Ankle isometric strength | Subjects were asked to test 1 time for 20 min before and after the intervention.
  Ankle dorsiflexion, plantarflexion, inversion and valgus isokinetic strengths were measured using the Humac Norm Multi-Joint Isokinetic Testing Instrument. Peak Torque (PT), Relative Peak Torque to Body Weight (PT/BW), and Total Work (TW) were measured during centripetal contraction at 60°/s and 180°/s angular velocities.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zheng, PhD, Principal Investigator — Tianjin University of Sport
Locations (1):
- Tianjin University of Sport, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No